CLINICAL TRIAL: NCT02995954
Title: Blood Pressure Reduction by Fixed-dose Compared to Free Dose Combination Therapy of ACE Inhibitor and Calcium Antagonist in Hypertensive Patients
Brief Title: Fixed vs Free Dose of ACEi/CCB Combination Therapy
Acronym: FixFree
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guido Iaccarino (Other)
Responsible Party: Sponsor-Investigator, Guido Iaccarino, Associate Professor of Internal of Medicine, Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona
Organization: Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iacca001
Record Dates: First submitted 2016-12-13; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Hypertension
Keywords: Combination therapy; ACE inhibitor Calcium Antagonist
MeSH Terms: conditions — Hypertension | interventions — amlodipine, perindopril drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed (Active Comparator): The Fixed group received one single tablet containing Perindopril/Amlodipine (Reaptan) at the appropriate dose
  Interventions: Drug: Perindopril/Amlodipine
- Free (Active Comparator): The Free group, received Perindopril and Amlodipine in separate tablets at the appropriate dose
  Interventions: Drug: Perindopril/Amlodipine

INTERVENTIONS:
Drug: Perindopril/Amlodipine — Single table containing Perindopril/Amlodipine
  Other Names: Perindopril amlodipine

SUMMARY:
The introduction of fixed combination of ACEi+CCB (Fixed) has significantly increased patients compliance and adherence to therapy. At the moment, however, there are no data suggesting the better control of once-daily fixed (Fixed) over free doses in separate administrations combination therapy in hypertensives.

In a population of 39 consecutive outpatient patients referred to the departmental Hypertension clinic of the University Hospital of Salerno Medical School with the first diagnosis of arterial hypertension, the investigators tested the hypothesis that the Fixed achieve a better control of blood pressure than the Free combination. Patients were randomized to either strategy and after 3 months patients underwent a clinical assessment to evaluate the antihypertensive effect.

DETAILED DESCRIPTION:
Study Population

Our study included 100 patients referred to the Hypertension Clinic of Salerno Medical School Hospital in Salerno, with the first diagnosis of arterial hypertension and in the absence of a previous treatment. At the time of enrollment visit, patients signed a consent to anonymous participation, in compliance with the regulations of good clinical practice and privacy. Study participants were 18-75 years old with essential hypertension (defined according to the ESH / ESC 2013 guidelines). Patients were excluded if patients had secondary hypertension, malignant hypertension, CRF (chronic renal failure), oncological conditions or cirrhosis. Patients were also excluded if patients had medical and surgical disorders that alter absorption, distribution, metabolism and excretion of drug treatment. The study protocol was approved by the competent University Hospital Ethical Committee.

Study Design

Patients were randomized to either fixed dose or free dose combination therapy, with Perindopril (5 or 10 mg) and Amlodipine (5 or 10 mg) with a 2:1 randomization design based on a power analysis. Doses were decided according to anthropometric, clinical, biochemical and instrumental doses by experienced medical staff. The Fixed group received one single tablet containing Perindopril/Amlodipine at the appropriate dose. The Free group, received Perindopril and Amlodipine in separate tablets at the appropriate dose. Groups were matched for age, sex, BMI, systolic BP (SBP) and diastolic BP (DBP). At baseline and at follow-up the investigators evaluated clinical (weight, height, BMI, heart rate, BP) and biochemical parameters (blood glucose, serum cholesterol, LDL, HDL, triglycerides, blood urea nitrogen, creatinine, creatinine clearance), as well as Electrocardiogram (ECG) and cardiac ultrasound.

Clinical parameters

In accordance with the ESH guidelines, BP assessment was carried out noting two measurements in the supine, in sitting and in standing position, spaced apart from 1-2 minutes. For the current study mean values in sitting position were considered. BP measurements were assessed by trained personnel using a dedicated, upper arm, electronic machine (Afib screen, Microlife, Italy) Anthropometric parameters.

The weight classes were defined by BMI [weight (kg)/height (m)2]. In adults, overweight is identified by a BMI of 25-29.9 kg/m2, and obesity by a BMI≥30 kg/m2.

Biochemical parameters

For each patient, the following laboratory tests were evaluated: fasting glucose, total cholesterol, LDL, HDL, triglycerides, blood urea nitrogen (BUN), serum creatinine and creatinine clearance (calculated with MDRD or Cockroft formula).

Fasting blood glucose greater than 126 mg/dl was used for screening for diabetes.

Follow-up with computerized medical records

The patient population was included in a central database that uses Wincare software (TSD-Projects, Milan, Italy), which contains separate electronic sheets for medical history, physical examination, laboratory tests, electrocardiogram, cardiac ultrasounds, other imaging tests and ambulatory blood pressure monitoring. The data was updated at each follow-up visit with a revaluation deadline set at three months. The data of each patient are stored on the hospital server and protected by a firewall system with password access.

Echocardiography

All patients were subjected to one-dimensional echocardiography (M-mode), two-dimensional (B-mode) and Doppler function via the 5-1MHz probe (E9, GE Healthcare).

Statistical analysis

Categorical data are presented as percent while continuous data are indicated as means ± standard error. The quantitative analysis was performed using T-test for unpaired data or ANOVA as appropriate, while the qualitative analysis was performed using non-parametric tests (χ2 test). A value of p-value <0.05 was considered statistically significant. All data were analyzed using Prism 6.0 (GraphPad Software, Inc., San Diego, CA).

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients with the first diagnosis of arterial hypertension and in the absence of a previous treatment.

Exclusion Criteria:

* Patients were excluded if patients had secondary hypertension, malignant hypertension, CRF (chronic renal failure), oncological conditions or cirrhosis.
* Patients were also excluded if patients had medical and surgical disorders that alter absorption, distribution, metabolism and excretion of drug treatment.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
systolic Blood pressure control | 3 months
  reduction in mmHg
Diastolic Blood pressure control | 3 months
  reduction in mmHg

SECONDARY OUTCOMES:
blood pressure control | 3 months
  percentage of patients with BP control

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni e Ruggi Hospital, Salerno, Salerno, Italy

IPD SHARING:
Plan to Share IPD: No